CLINICAL TRIAL: NCT06330194
Title: Glucose Control With a Next Generation Advanced Insulin Delivery System in Adults With Diabetes and Advanced Renal Disease
Brief Title: Next Generation Advanced Insulin Delivery System in Adults With Diabetes and Advanced Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tobias Bomholt, Tobias Bomholt, MD, PhD, Post.doc., Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AID-study
Record Dates: First submitted 2024-02-20; First posted 2024-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dialysis; Chronic Kidney Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Hemodialysis; Peritoneal Dialysis
Keywords: Insulin Infusion Systems; Continuous Glucose Monitoring; Randomized Controlled Trial; Equipment Safety; Glycemic Control; Time-in-range
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Insemination, Artificial, Heterologous; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Design: Prospective, open-label, two-stage randomised-crossover study.
  Population: Patients with type 1 or type 2 diabetes undergoing hemodialysis (n=5), peritoneal dialysis (n=5) or chronic kidney disease stage 3b to stage 5 (n=5).
  Methods: Participants entering the study will have a four-to-six-week run-in phase with diabetes education. During the run-in phase three weeks of unblinded continous glucose monitoring (CGM) will be performed to assess baseline glucose levels.
  All participants will be randomized to receive either eight weeks with an advanced insulin delivery (AID) System or eight weeks of control (usual care) with cross over at the end of the first eight weeks.
  CGM study outcome data will be collected by identical methods, using unblinded-CGM devices, for participants in both intervention and control study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): 2nd Generation Automated Insulin Delivery system (Medtronic MiniMed 780G)
  Interventions: Device: 2nd Generation Automated Insulin Delivery (AID) system
- Control Group (No Intervention): Usual care consisting of participants current insulin-treatment (either multiple daily injection with insulin or traditional insulin pump therapy with manual determination of insulin dosing) and real-time CGM if already used.

INTERVENTIONS:
Device: 2nd Generation Automated Insulin Delivery (AID) system — The AID system will initially commence delivery by insulin pump post-randomisation without the AID in operation and with predictive low glucose suspend activated for a period of two weeks. Once safety has been established, the autocorrect function can be activated and the setpoint reduced to 5.5 mmol/L. Throughout the study insulin pump uploads will be reviewed twice weekly initially and at least weekly thereafter.
  Other Names: Medtronic MiniMed 780G
  Arms: Intervention Group

SUMMARY:
The goal of this this randomized, clinical trial is to test an automated insulin delivery system (AID) in people with type 1 or type 2 diabetes who are on hemodialysis, peritoneal dialysis, or have advanced chronic kidney disease (CKD).

The main objective is:

• To test if the AID is superior in regulating blood sugar levels compared with usual care in patients with advanced renal disease

Secondary objectives are:

• To evaluate the impact on life quality, incidence of low blood sugar, and if the treatment is feasible in this population

Participants will be randomized to receive either eight weeks with the AID System (780G from Medtronic) or eight weeks of Control (usual care) with cross over at the end of the first eight weeks.

Researchers will compare blood sugar levels between the AID group and the Control group to determine if the AID system is superior in regulating blood sugar levels.

DETAILED DESCRIPTION:
Dialysis patients with diabetes have a very short life expectancy likely caused by a high incidence of co-morbidities combined with an increased risk of hypoglycaemia and poor glycaemic control. In the past decades various diabetes technologies have revolutionised treatment, primarily in type 1 diabetes, but have also shown effect in type 2 diabetes. The Automated Insulin Delivery (AID) system combines continuous glucose monitoring (CGM) with an insulin pump that automatically infuse short-acting insulin subcutaneously and has shown remarkable results in improving glucose levels. We hypothesise that the AID system can lead to a substantial improvement in glycaemic control for patients receiving haemodialysis (HD), peritoneal dialysis (PD) and patients with chronic kidney disease (CKD) stage 3b to 5 (not on dialysis).

The primary objective is to determine if the AID system is superior in regulating glucose levels, in people living with type 1 and type 2 diabetes, receiving HD, PD or having advanced CKD, compared with usual care. Secondary objectives are to evaluate the impact on life quality, incidence of hypoglycaemia and if this treatment is feasible for this population

This prospective, open-label, two-stage randomized-crossover study is conducted at the Department of Nephrology, Rigshospitalet Copenhagen and Steno Diabetes Center Copenhagen. The study is performed in collaboration with six Australian centres (St Vincent's Melbourne, Royal Melbourne, Austin, Cairns Base, Flinders, and Canberra Hospitals).

A total of 15 participants will be recruited in Copenhagen, with participants evenly distributed across the three disease categories (HD, PD, and advanced CKD). Data collected from Copenhagen will be pooled with data obtained from the Australian centers.

Participants entering the study will have a four-to-six-week run-in phase with diabetes education (carbohydrate counting, inserting of CGM etc). Training will consist of three sessions of 2-4 hours with a dedicated diabetes nurse. During the run-in phase three weeks of unblinded CGM will be performed to assess baseline glucose levels. All participants will be randomized 1:1 to receive either eight weeks with the AID System (780G from Medtronic) or eight weeks of control (usual care) with cross over at the end of the first eight weeks.

The trial will be conducted in compliance with the Good Clinical Practice (GCP) guidelines, and written informed consent will be obtained before any trial activities are performed. The project including a plan for the handling of personal information will be approved by the Danish Data Protection Agency before initiation. If necessary, the Danish Medicines Agency and the responsible GCP unit will be granted access to journals, documents, and other materials relevant to the project. All participants will be assigned with a subject number and will be recorded on data sheets. Only tubes will appear with subject number and trial ID. Information on full name and social security and subject numbers will be stored separately.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial-related procedures are performed
2. Type 1 diabetes of at least 1-year duration or insulin requiring type 2 diabetes (Total insulin dose should be below 200 IE per day)
3. Maintenance HD, PD, or CKD stage 3b-5 (not on dialysis).
4. Subject must be willing and able to comply with trial protocol
5. HbA1c <91 mmol/mol (10.5%)

All participants will require to have internet or mobile phone access enabling upload of the AID system data to cloud based software.

Exclusion Criteria:

1. History of ketoacidosis within the past 6 months
2. Moderate to severe cognitive impairment
3. Major allergy to tape/ adhesives
4. Women who are pregnant or planning pregnancy
5. Life-expectancy to <6 months
6. Major psychiatric history
7. Treatment with sulphonylureas in pre-dialysis participants (SGLT2 inhibitors, metformin, and GLP1 analogues may be used within regulatory guidelines)
8. Treatment with non-insulin glucose lowering therapies may not be used on dialysis participants (with the exception of GLP1 agonists used in preparation for transplantation)
9. Systemic steroid treatment within 4 weeks (stable doses of steroids >8 weeks allowed)
10. Visual impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Percent time in sensor glucose target range (3.9-10.0 mmol/L) | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM

SECONDARY OUTCOMES:
Proportion of time spent <2.8 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent <3.0 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent <3.3 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent <3.9 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent 3.9-7.8 | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent >10.0 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent >13.9 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Proportion of time spent >16.7 mmol/L | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Glucose variability (SD and coefficient of variation) | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Mean glucose | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
HbA1c | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Blood sample
Episodes of CGM time in < 3.0 mmol/L range lasting >15 minutes | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Assessed by 3 continuous weeks of CGM
Diabetic ketoacidosis og Hyperosmolar non-ketotic hyperglycemia | Week 0-22
  Hospital presentations with either of the above
eGFR (estimated glomerular filtration rate) | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Based on serum creatinine measurements, using the CKD-EPI equation. Only measured in patients from the CKD-group
Potassium pre-dialysis | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Blood sample. Only measured in patients from the HD-group
Urine albumine-to-creatinine ratio | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Urine sample. Only measured in patients from the CKD-group
Actigraph Metrics for sleep architecture | End of run in phase: week 3-5; end of phase 1: week 11-13; end of phase 2: week 20-22
  Used concurrently with the CGM
Sleep diary | Week 6-22
Proportion of time Automode is active | Weekly assessed: week 6-22
  Registered through uploads from insulin pump in the intervention arm
Diabetic ketoacidosis | Week 0-22
Severe hypoglycemia | Week 0-22
  Requiring third party assistance
Serious Adverse Event | Week 0-22
Unanticipated Serious Adverse Device Event | Week 0-22
Satisfaction with diabetes treatment | Enrollment visit: week 0; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: The Diabetes Treatment Satisfaction Questionnaire status [DTSQs]
Satisfaction with diabetes treatment | End of phase 1: week 14; end of phase 2: week 22
  Questionnaire: The Diabetes Treatment Satisfaction Questionnaire control version [DTSQc]
Fear of hypoglycaemia | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: Hypoglycaemia Fear Survey [HFS-II]
Hypoglycaemia awareness | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: Gold Score and Clarke Score
Diabetes distress | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: Problem Areas in Diabetes [PAID]
Sleep Quality | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: Pittsburgh Sleep Quality Index [PSQI]
Cognitive function | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: Montreal Cognitive Assessment (MOCA)
Sarcopenia | End of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  SARC-F questionnaire
Semi-structured interview | End of phase 1: week 14; end of phase 2: week 22
  Influence of kidney disease on diabetes management and experience with the AID. Only performed in intervention arm.
Health-related quality of life | Enrollment visit: week 0; end of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: EQ-5D
Frailty | End of run in phase: week 6; end of phase 1: week 14; end of phase 2: week 22
  Questionnaire: Fried Frailty

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Bomholt, MD, PhD, Principal Investigator — Department of Nephrology, Rigshospitalet, University of Copenhagen
Locations (1):
- Tobias Bomholt, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No